CLINICAL TRIAL: NCT05054738
Title: Impact of Combined Recovery Program and Home Telehealth Among Veterans With Substance Use Disorders in the VA Inpatient Setting
Brief Title: CRP and S&A for Inpatient Veterans
Acronym: CRP and S&A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 19-395
Record Dates: First submitted 2021-09-02; First posted 2021-09-23 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Alcoholism; Substance-related Disorders; Dual Diagnosis
Keywords: Alcoholism; Substance-related disorders; Dual Diagnosis
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Between groups randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI and research staff providing follow up assessments will be blinded to participants study condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Combined Recovery Program (CRP)+Treatment-as-usual (TAU) (Experimental): Combined Recovery Program (CRP) is a six-session motivational enhancement and daily living skills therapy workshop provided while on the inpatient unit. Attendance of CRP will be in addition to Treatment as Usual (TAU), that is, standard inpatient programming.
  Interventions: Behavioral: Combined Recovery Program
- CRP+ Stable & Able (S&A)+TAU (Active Comparator): Combined Recovery Program (CRP) a six-session motivational enhancement and daily living skills therapy workshop provided while on the inpatient unit, plus a home telehealth program (Stable & Able) which begins on day 1 of hospital discharge. Attendance of CRP and S&A will be in addition to TAU, that is, standard inpatient programming.
  Interventions: Behavioral: Combined Recovery Program; Behavioral: Stable & Able (S&A)
- Treatment-as-usual only (TAU): (No Intervention): TAU will only receive the usual care on the inpatient unit including medical and medication management.

INTERVENTIONS:
Behavioral: Combined Recovery Program — A six-session treatment group designed to explore goals, values, and personal strengths about making a change for overall quality of life, health and well-being combined with skill building designed for helping to live a more stable life in their own home that will include money management for financial success and home maintenance.
  Arms: CRP+ Stable & Able (S&A)+TAU; Combined Recovery Program (CRP)+Treatment-as-usual (TAU)
Behavioral: Stable & Able (S&A) — A 90-day Home Telehealth program designed to help maintain skills to stay sober.
  Arms: CRP+ Stable & Able (S&A)+TAU

SUMMARY:
The purpose of this study is to evaluate how well three types of treatments work to improve the outcomes for people with substance use problems. Veterans admitted to the Charleston VA Psychiatric inpatient unit may be invited to participate. The three types of treatments that will be evaluated are:

1. Combined Recovery Program (CRP), a six-session treatment group delivered on the inpatient unit.
2. A Home Telehealth program, called Stable and Able (S&A), provided just prior to discharge and provides additional support for up to 3 months
3. Treatment-as-usual (TAU), which is the treatment currently provided on the unit, consisting of various mental health topics and sessions designed to help with recovery.

Participation begins on the inpatient unit, beginning with CRP and/or TAU, and may continue with S&A post discharge. Participants will be followed up at 1 and 3- months post treatment.

DETAILED DESCRIPTION:
Background:

High inpatient readmissions among Veterans with substance use disorders (SUD) constitutes a costly and persistent healthcare problem. Studies demonstrate that patients with SUDs return to inpatient treatment multiple times and that high inpatient service utilization in this population is associated with high rates of co-occurring mental illness (SUD/MI), homelessness, suicidality, and continued impairment in health and social functioning. A significant proportion (21%) of Veterans with SUD/MI are homeless, at high-risk for suicide, and represent one of the largest, most chronic groups of psychiatric patients treated in the VA Healthcare System. In effort to ameliorate inpatient readmission rates, VHA Handbook 1160.06, drafted in 2013, espouses the development and implementation of uniform recovery-oriented mental health (MH) services, which include treatment of SUDs addressing goals of recovery, improved quality of life, and community integration. The three types of treatments that will be evaluated are:

1. Combined Recovery Program (CRP), a six-session treatment group designed to explore goals, values, and personal strengths about making a change for overall quality of life, health and well-being combined with skill building designed for helping to live a more stable life in their own home that will include money management for financial success and home maintenance.
2. A Home Telehealth program, called Stable and Able (S&A), designed to help maintain skills to stay sober and allows continued communication with one of the mental health staff on a daily basis to provide additional support for the next 3 months after discharge.
3. Treatment-as-usual (TAU), which is the treatment currently provided on the unit, consisting of various mental health topics and sessions designed to help with recovery.

All participant will receive TAU.

Objectives:

Specific Aim I: Assess the relative effects of Treatment Engagement and Substance Use [and SUD-related problems] between CRP+S&A+TAU vs. CRP+TAU and CRP+S&A+TAU vs. TAU only by 3-mos follow-up.

Primary Hypothesis 1a: Treatment Engagement: Participants in CRP + S&A+TAU will attend more outpatient SUD treatment sessions and general MH treatment sessions compared to participants in CRP and to TAU.

Primary Hypothesis 1b: Substance Use: Participants in CRP + S&A+TAU will lower quantity and frequency of substance use and SUD-related problems compared to participants in CRP+TAU and to TAU only.

Secondary Hypothesis 1c: Preventable Services: Participants in CRP + S&A+TAU will reduce Preventable Healthcare Services (hospital readmissions and emergency department visits) compared to participants in CRP+TAU and to TAU only.

Secondary Hypothesis 1d: Participants in CRP + S&A+TAU will report Greater QoL; # of Days Living in Stable Housing; and # of Days Engaging in Community Events and/or Activities compared to CRP+TAU and to TAU only.

Specific Aim II: Conduct Veteran participant and Staff thematic interviews and to assess qualitative facilitators and barriers to implementation.

Methods:

195 Veterans with SUDs admitted into the Charleston VAMC inpatient unit will be recruited. Participants will be randomly assigned to: (1) CRP + S&A + TAU; (2) CRP+TAU; and (3) TAU. All participants will be followed-up at 1 and 3-months and data analyzed using mixed methods.

ELIGIBILITY:
Inclusion Criteria:

* Meeting DSM-V criteria for current SUD diagnosis of alcohol and/or illicit drug use disorder
* Use of substances in past 30 days prior to date of index inpatient admission
* Able to comprehend English
* Able to provide informed consent
* Functioning at an intellectual level sufficient to allow accurate completion of all assessments
* Willing to commit to 6 group inpatient therapy sessions, telehealth S&A, as well as baseline, and 1-and 3-month follow-up assessments

Exclusion Criteria:

* Auditory or visual impairment that would interfere with study procedures
* Inability to speak or understand English
* Acutely psychotic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Standard Ethanol Content Units (SECs) Baseline | Baseline
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol at Baseline (e.g., the past 30 days is defined as 'Baseline'). Amount of alcohol consumption was converted to standard ethanol content units (SECs; or standard drinks) equivalent to 0.5 oz. of ethanol. This measure represents ALL standard drinks consumed within the stated time period.
Standard Ethanol Content Units (SECs) at 1 month | 1 month
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days after the first day of treatment. Amount of alcohol consumption was converted to standard ethanol content units (SECs; or standard drinks) equivalent to 0.5 oz. of ethanol. This measure represents ALL standard drinks consumed within the stated time period.
Standard Ethanol Content Units (SECs) at 3 month | 3 Month
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 60 days after the 1-month follow-up. Amount of alcohol consumption was converted to standard ethanol content units (SECs; or standard drinks) equivalent to 0.5 oz. of ethanol. This measure represents ALL standard drinks consumed within the stated time period.
Peak SEC at Baseline | Baseline
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days prior to baseline. Amount of alcohol consumption was converted to standard ethanol content units (SECs; or standard drinks) equivalent to 0.5 oz. of ethanol. This measure represents the most standard drinks consumed in a single day within the stated time period.
Peak at 1 Month | 30 days
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days after the first day of treatment. Amount of alcohol consumption was converted to standard ethanol content units (SECs; or standard drinks) equivalent to 0.5 oz. of ethanol. This measure represents the most standard drinks consumed in a single day within the stated time period.
Peak at 3 Month | 3 Month
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 60 days after the 1-month follow-up. Amount of alcohol consumption was converted to standard ethanol content units (SECs; or standard drinks) equivalent to 0.5 oz. of ethanol. This measure represents the most standard drinks consumed in a single day within the stated time period.
Alcohol Drink Days at Baseline | Baseline
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days prior to Baseline. This measure represents the number of days any alcohol was consumed within the stated time period.
Alcohol Drink Days at 1 Month | 30 days
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days after the first day of treatment. This measure represents the number of days any alcohol was consumed within the stated time period.
Alcohol Drink Days at 3 Month | 3 Month
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 60 days after the 1-month follow-up. This measure represents the number of days any alcohol was consumed within the stated time period.
Binge Drink Days at Baseline | Baseline
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days prior to Baseline. This measure represents the number of days the participant binge drank.
Binge Drink Days at 1 month | 1 month
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days after the first day of treatment. This measure represents the number of days the participant binge drank within the stated time period.
Binge Drink Days at 3 Month | 3 month
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 60 days after the 1-month follow-up. This measure represents the number of days the participant binge drank within the stated time period.
Illicit Drug Use Days at Baseline | Baseline
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of drug use in the 30 days prior to Baseline. This measure represents the number of illicit drug use days within the stated time period.
Illicit Drug Use Days at 1 Month | 30 days
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of drug use in the 30 days after the first day of treatment. This measure represents the number of illicit drug use days within the stated time period.
Illicit Drug Use Days at 3 month | 3 Month
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of drug use in the 60 days after the 1-month follow-up. This measure represents the number of illicit drug use days within the stated time period.
Substance Use Disorder Treatment Sessions at Baseline | Baseline
  A Treatment Attendance Calendar was used to record the number of objective treatment sessions documented in each participants VA Electronic Health Record System for the 30 days prior to Baseline. Treatment sessions included the outpatient substance use disorder treatment group sessions and individual sessions.
Substance Use Disorder Treatment Sessions at 1 month | 30 days
  A Treatment Attendance Calendar was used to record the number of objective treatment sessions documented in each participants VA Electronic Health Record System for the 30 days after the first day of treatment. Treatment sessions included the outpatient substance use disorder treatment group sessions and individual sessions.
Substance Use Disorder Treatment Sessions at 3 Month | 3 Month
  A Treatment Attendance Calendar was used to record the number of objective treatment sessions documented in each participants VA Electronic Health Record System for the 30 days after the 1-month follow-up. Treatment sessions included the outpatient substance use disorder treatment group sessions and individual sessions.
Twelve-Step Sessions Attended at Baseline | Baseline
  A Treatment Attendance Calendar was used to record the number of self-reported 12-step sessions attended 30 days prior to Baseline.
Twelve-Step Sessions Attended at 1 Month | 30 days
  A Treatment Attendance Calendar was used to record the number of self-reported 12-step sessions attended 30 days after the first day of treatment.
Twelve-Step Sessions Attended at 3 month | 3 Month
  A Treatment Attendance Calendar was used to record the number of self-reported 12-step sessions attended 60 days after the 1-month follow-up.
Community Participation Activities at Baseline | Baseline
  A calendar was used to record the number of times a participant participated in an activity in the community (e.g. museum, library, baseball game) in the 30 days prior to Baseline.
Community Participation Activities at 1 month | 30 days
  A calendar was used to record the number of times a participant participated in an activity in the community (e.g. museum, library, baseball game) in the 30 days after the 1st day of treatment.
Community Participation Activities at 3 month | 3 Month
  A calendar was used to record the number of times a participant participated in an activity in the community (e.g. museum, library, baseball game)in the 60 days after the 1-month follow-up.
Mental Health Treatment Sessions at Baseline | Baseline
  A Treatment Attendance Calendar was used to record the number of objective treatment sessions documented in each participants VA Computerized Patient Record System for the 30 days prior to Baseline. Treatment sessions included individual sessions with outpatient mental health staff.
Mental Health Treatment Sessions at 1 month | 30 days
  A Treatment Attendance Calendar was used to record the number of objective treatment sessions documented in each participants VA Computerized Patient Record System for the 30 days after discharge. Treatment sessions included individual sessions with outpatient mental health staff.
Mental Health Treatment Sessions at 3 month | 3 Month
  A Treatment Attendance Calendar was used to record the number of objective treatment sessions documented in each participants VA Computerized Patient Record System for the 60 days after the 1-month follow-up. Treatment sessions included individual sessions with outpatient mental health staff.

SECONDARY OUTCOMES:
Addiction Severity Index-Lite (ASI-Lite) at Baseline for Alcohol Use | Baseline
  The ASI-Lite will be used to measure addiction severity Min value:0 Max value: 1 Higher score indicates greater problem severity
Addiction Severity Index-Lite (ASI-Lite) at 1 month for Alcohol Use | 30 days
  The ASI-Lite will be used to measure addiction severity Min value:0 Max value: 1 Higher score indicates greater problem severity
Addiction Severity Index-Lite (ASI-Lite) at 3 month for Alcohol Use | 3 Month
  The ASI-Lite will be used to measure addiction severity Min value:0 Max value: 1 Higher score indicates greater problem severity
Addiction Severity Index-Lite (ASI-Lite) at Baseline for Psychiatric Status | Baseline
  The ASI-Lite will be used to measure addiction severity Min value:0 Max value: 1 Higher score indicates greater problem severity
Addiction Severity Index-Lite (ASI-Lite) at 1 month for Psychiatric Status | 30 days
  The ASI-Lite will be used to measure addiction severity Min value:0 Max value: 1 Higher score indicates greater problem severity
Addiction Severity Index-Lite (ASI-Lite) at 3 month for Psychiatric Status | 3 Month
  The ASI-Lite will be used to measure addiction severity Min value:0 Max value: 1 Higher score indicates greater problem severity
Short Inventory of Problems (SIP) at Baseline | Baseline
  Min value:0 Max value: 45 Higher score indicates higher number of consequences from alcohol and drug use
Short Inventory of Problems (SIP) at 1 month | 30 days
  Min value:0 Max value: 45 Higher score indicates higher number of consequences from alcohol and drug use
Short Inventory of Problems (SIP) at 3 month | 3 Month
  Min value:0 Max value: 45 Higher score indicates higher number of consequences from alcohol and drug use
Quality of Life Survey (QOLS) at Baseline | Baseline
  Min value:16 Max value:112 Higher score indicates higher quality of life
Quality of Life Survey (QOLS) at 1 month | 30 days
  Min value:16 Max value:112 Higher score indicates higher quality of life
Quality of Life Survey (QOLS) at 3 month | 3 Month
  Min value:16 Max value:112 Higher score indicates higher quality of life
Brief Symptom Inventory (BSI-18) at Baseline | Baseline
  Min value:0 Max value:72 Higher score indicates higher psychological distress
Brief Symptom Inventory (BSI-18) at 1 month | 30 days
  Min value:0 Max value:72 Higher score indicates higher psychological distress
Brief Symptom Inventory (BSI-18) at 3 month | 3 Month
  Min value:0 Max value:72 Higher score indicates higher psychological distress
Treatment Motivation Questionnaire (TMQ) at Baseline | Baseline
  The TMQ will be used to measure self-reported interest in attending treatment Scores within each subscale are averaged
  External:
  Min value:1 Max value:7 External: Higher score indicates higher external reasons for attending treatment (e.g. referred to treatment by legal system)
  Internal:
  Min value:1 Max value:7 Internal: Higher score indicates higher internal reasons for attending treatment (e.g. personal choice to attend treatment)
Treatment Motivation Questionnaire (TMQ) at 1 month | 30 days
  The TMQ will be used to measure self-reported interest in attending treatment Scores within each subscale are averaged
  External:
  Min value:1 Max value:7 External: Higher score indicates higher external reasons for attending treatment (e.g. referred to treatment by legal system)
  Internal:
  Min value:1 Max value:7 Internal: Higher score indicates higher internal reasons for attending treatment (e.g. personal choice to attend treatment)
Treatment Motivation Questionnaire (TMQ) at 3 month | 3 Month
  The TMQ will be used to measure self-reported interest in attending treatment Scores within each subscale are averaged
  External:
  Min value:1 Max value:7 External: Higher score indicates higher external reasons for attending treatment (e.g. referred to treatment by legal system)
  Internal:
  Min value:1 Max value:7 Internal: Higher score indicates higher internal reasons for attending treatment (e.g. personal choice to attend treatment)
Fagerstrom Test for Nicotine Dependence at Baseline | Baseline
  Min:0 Max:10 Higher score indicates higher level of nicotine dependence
Preventable Healthcare Services at 1 month Baseline | 30 days
  A Treatment Attendance Calendar was used to record the number of separate psychiatric inpatient admissions and emergency department visits documented in each participants VA Computerized Patient Record System for the 30 days prior to Baseline.
Preventable Healthcare Services at 1 month | 30 days
  A Treatment Attendance Calendar was used to record the number of separate psychiatric inpatient admissions and emergency department visits documented in each participants VA Computerized Patient Record System for the 30 days after discharge.
Preventable Healthcare Services at 3 month | 3 Month
  A Treatment Attendance Calendar was used to record the number of separate psychiatric inpatient admissions and emergency department visits documented in each participants VA Computerized Patient Record System for the 60 days after the 1-month follow-up.
Housing Status Inventory at Baseline | Baseline
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of housing status for the 30 days prior to Baseline.
Housing Status Inventory at 1 month | 30 days
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of housing status for the 30 days after discharge.
Housing Status Inventory at 3 month | 3 Month
  The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of housing status for the 60 days after the 1-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J. Santa Ana, PhD MA BA, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No